CLINICAL TRIAL: NCT01854073
Title: Use of Hyoscine Butyl Bromide for Management of Prolonged Labor in Nulliparous Women, A Randomized Controlled Trial
Brief Title: Hyoscine Butyl Bromide for Management of Prolonged Labor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Armed Forces Hospitals, Southern Region, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Mohamed Ellaithy, Assistant professor of Obstetrics & Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AFHSR-5-2013
Record Dates: First submitted 2013-05-11; First posted 2013-05-15 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Prolonged Labor
MeSH Terms: interventions — Butylscopolammonium Bromide; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Group A, will receive injection Hyoscine butyl bromide 20 mg first dose at the time of amniotomy, and second dose 2 hours after.
  Interventions: Drug: Hyoscine butyl bromide
- Group B (Placebo Comparator): Group B, will receive normal saline same volume first dose at the time of amniotomy, and second dose 2 hours after.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Hyoscine butyl bromide
  Other Names: Buscopan
  Arms: Group A
Drug: Normal saline
  Other Names: Sodium chloride 0.9%
  Arms: Group B

SUMMARY:
To determine the value of using Hyoscine as an antispasmodic drug for the management of prolonged labor in nulliparous women at term.

DETAILED DESCRIPTION:
Management of prolonged labor represents a challenging area in the daily obstetric practice. In 1993, Handa and Laros defined the arrest of active phase of labor, as failure of labor progress for 2 hours or more, and in 1994, WHO has proposed labor management partograph in which protraction is defined as < 1cm/hour cervical dilatation for a minimum of 4 hours.

Prolong labor increase the risks of maternal exhaustion, postpartum hemorrhage, sepsis, fetal distress and admission to the neonatal intensive care unit. The treatment of prolonged labor is highly desirable goal of intrapartum care, both from prospective of maternal and fetal wellbeing and for the provider of the birth services. Management of prolonged labor entails shorter exposure to pain, anxiety, and stress, and would thus translate into a major improvement in maternal satisfaction with child birth experience.

Several methods have been used for management of prolonged labor including amniotomy and oxytocin. Amniotomy can cause infection, and can be combined with oxytocin for better results while oxytocin can cause uterine hyper stimulation, water intoxication, vomiting, diarrhea, fetal distress, and neonatal jaundice.

Use of antispasmodics for reducing the duration of labor was first described in 1937 by Hirsch, who reported a decrease in labor length by two to four hours following intrapartum administration of an antispasmodic like drug (Syntropan®), mainly among older nulliparous, this was followed by many studies that investigated the role of antispasmodics in prevention of prolonged labor, however none of the these studies assessed the value of the antispasmodic for the treatment of prolonged labor; a recent Cochrane review advised that a rigorously designed well conducted randomized controlled trial with a large sample size would be beneficial to answer the question.

Hyoscine butyl bromide is spasmolytic drug that act by competitive antagonism to acetyl choline at post ganglionic parasympathetic nerve ending. It is claimed to reduce duration of labor by accelerating cervical dilatation without major side effects. It reduces the spasm of the smooth muscles. Although the efficacy of Hyoscine has been proven in various studies there is no clear evidence to recommend their routine use in management of prolonged labor.

The objective of the current study is to determine the use of Hyoscine as an antispasmodic drug for the management of prolonged labor in nulliparous women at term, managed according to a standard intrapartum protocol.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women.
* Prolonged labor defined as no progress of labor for 2 hours or more.
* Gestational age ≥ 37 weeks.
* Singleton pregnancy.
* Cephalic presentation.
* Cervical dilatation ≥ 5 cm.
* Intact fetal membranes.
* No evidence of maternal or fetal distress.
* Average size baby.

Exclusion Criteria:

* Multigravid women.
* Multifetal pregnancy.
* History of cervical surgery.
* Blood pressure > 150/90 mmHg.
* Mal-presentation and mal-positions.
* Hypersensitivity to Hyoscine.
* Contraindication for vaginal delivery.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Caesarean section rate for failure to progress | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ellaithy, MD, Principal Investigator — Ain Shams University
Locations (1):
- Labor and delivery ward of Armed Forces Hospital, Southern Region., Khamis Mushait, 'Asir Region, Saudi Arabia